CLINICAL TRIAL: NCT00324285
Title: Oral Rehydration SolutionContaining Amylase Resistant Starch in Severely Malnourished Children With Watery Diarrhoea Due to Vibrio Cholerae
Brief Title: Oral Rehydration SolutionContaining Amylase Resistant Starch in Severely Malnourished Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001-007
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2006-05

CONDITIONS: Diarrhoea; Severe Malnutrition
Keywords: Diarrhoea; severe malnutrition; amylase resistant starch; ORS
MeSH Terms: conditions — Diarrhea; Malnutrition

INTERVENTIONS:
Drug: Amylase resistant starch added ORS

SUMMARY:
Severe malnutrition is associated with a high rate of mortality, even when using the latest WHO recommendations. Watery diarrhea as observed in cholera is an additional vital risk to those children. The fragility of the children together with the complexity of the pathophysiology and the simplicity of the medical environment where the treatment is delivered are serious constraints for the development of new therapies. Dehydration is a special immediate risk in those children who already displayed altered body distribution of water with potassium, magnesium, zinc and other nutrient deficiency. Dehydration is also often associated with a decrease in appetite. In addition, the intestinal function is altered both by the infectious agent and the nutritional status of the child. Recommended therapy for those children comprises oral rehydration with ReSoMaL (modified ORS for use in severely malnourished children recommended by WHO), at a relatively low rate, with permanent monitoring; in addition, breastfeeding should not be interrupted and feeding with F100 (Milk based formula diet for use in severely malnourished children recommended by WHO) is recommended. Recently, amylase-resistant starch added to a standard WHO-ORS has been shown to reduce the duration and severity of adults with cholera. The rationale for using amylase-resistant starch was that when starch enters the colon it is metabolized by the bacteria. The short-chain fatty acids thus produced stimulate sodium absorption in the colon, just like glucose stimulates water absorption in the small intestine. In addition, this treatment would be of particular interest in malnutrition because short-chain fatty acids are specific energetic substrate for the colon.In the present project, we propose to test the hypothesis that addition of amylase-resistant starch to the already recommended treatment of severely malnourished children with cholera reduces the severity and duration of diarrhea; this could be achieved through the effect of short-chain fatty acids on colonic sodium absorption. In addition, a better recovery from malnutrition could be achieved through the energy provided by short-chain fatty acids to the colon and improved appetite through improved rehydration. Thus, the aim of the study is to measure the effect of amylase-resistant starch added to an already accepted treatment (with minimal changes) at the rehydration and rehabilitation phases of the treatment. A total of 210 children aged 6 mo to 60 mo will be studied in three groups : a) glucose based ORS and amylase-resistant starch; b) glucose based ORS without amylase resistant starch ; c) rice based ORS . The major outcome variables on the first phase (diarrhoeal duration and stool output), and second phase (food intake, weight gain) will be compared between the two treatment groups. The result of the study if found effective in reducing the duration of diarrhoea, enhance recovery from diarrhoea and malnutrition in severely malnourished children, will contribute to better case management of these children.

DETAILED DESCRIPTION:
STUDY DESIGN This is a randomized controlled clinical trial.

Subjects

Inclusion criteria:

1. History of acute watery diarrhoea of <72 hrs.
2. Either sex.
3. Age - 6m to 60 months
4. Some or severe dehydration.
5. Wt for Ht <70% of NCHS median: with or without edema.
6. Dark field examination positive for Vibrio cholerae.
7. Consent given by the patient or legal guardian.

Exclusion criteria:

1. Bloody diarrhoea.
2. Severe infection (e.g. severe pneumonia, clinical sepsis, meningitis).
3. Those who received antibiotics/antimicrobial for the current illness Sample Size Sample size is calculated on the basis of duration of diarrhoea of recently completed study with WHO-ORS vs. ReSoMaL in severely malnourished children with diarrhoea (65±46 vs. 61±45). Expecting 35% reduction of duration of diarrhoea with the proposed new treatment considering 5% level of significance and 80% power, the sample size in each group is 70. Considering the stool weight, with reference of (stool wt. 158±95 when treated with WHO ORS) in severely malnourished children with cholera, the sample size was estimated to be 65 in each group, expecting 30% reduction in stool weight during the first 24 hours with the new treatment and considering 5% level of significance and 80% power. Finally we consider to study 70 patients in each treatment group.

Randomization

After enrollment into the study the patients will be randomized to receive one of the following three solutions:

1. Modified glucose based WHO ORS
2. Modified glucose WHO ORS plus 50 g/L amylase resistant starch.
3. Modified rice based ORS

Since a significant proportion of children might present with ALRI, randomization will be stratified into two strata:

1. Children with ALRI
2. Children without ALRI Accordingly, two randomization list will be prepared. The randomization list will be prepared using random table of permuted block of variable length.

   Baseline information

   A baseline history and examination will be obtained in order to:

   4determine the subject's eligibility for inclusion in the study; 4collect the relevant data prior to beginning the study.

   The baseline history and examination will include:

   4identification of the patient; 4a description of the symptoms prior to admission and their duration; 4detail of any treatment given for the illness before admission; 4results of physical examination including the state of hydration.

   Assessment of dehydration This will be done according to the modified WHO guideline used in ICDDR,B. (Appendix-III).

   Laboratory tests After admission blood for Hct, total protein, glucose, and serum electrolytes will be sent before initiation of the assigned ORS. Serum electrolytes will be repeated after 24 and 48 hours after initiation of ORS therapy. Stool sample will be sent for microscopy (including cryptosporidium and giardia) and culture for shigella, salmonella, Vibrio cholerae and ELISA for rotavirus will be done. Other relevant investigations like Total WBC count, Differential count and urine microscopy will be done routinely. Chest X-ray and/or Blood culture will be done, if necessary.

   For all blood tests 3 ml of blood will be drawn from a suitable vein in the hand.

   Estimation of fecal Starch and SCFAs Feces from 50 patients will be collected in buckets. The first 24 h collected feces will be weighed and aliquot will be taken and stored at -20o C until the analysis of SCFAs by HPLC. The second and third stool samples will be collected from 24-48 h and 48-72 h respectively. The feces will be weighed and aliquot will be stored at -20oC for the determination of SCFAs.

   Fecal starch will be measured enzymatically with a starch-assay kit (Total Starch Assay Procedure, Megazyme, Warriewood, Australia).

   Case Management (Acute Phase) After randomization the children will be treated following the standardized protocol for management of severely malnourished children used at ICDDR,B hospital (2,12).

   Fluid Therapy (oral) Dehydration assessment will be done according to the WHO guideline modified for in our last multicentre clinical trial of reduced osmolarity ORS in adult cholera and children with watery diarrhoea (17). In children with some dehydration, the fluid deficit will be corrected with the assigned ORS @ 10 ml/kg/hour for the first two hours, then 5 ml/kg/hour until the deficit will be corrected. In addition, on going stool losses will be corrected @ 5-10 ml/kg/ after each watery stool. For high purging patient, the ORS intake will be adjusted according to the on going stool loss. ORS therapy will be continued until diarrhoea ceased. Randomization of patient, taking consent and darkfield report collection will not take more than 20 minutes. If delayed more than 20 minutes the children will be offered glucose based ORS and subsequently switched over to the assigned ORS. Children with severe dehydration, initial rehydration will be done with IV fluid (cholera saline; Na 133 mmol/L, Cl 98 mmol/L, K 13 mmol/L and Acetate equivalent to HCO3 48 mmol/ L) until the patient is out of shock or disappearance of signs of severe dehydration then the rest of rehydration will be done as for rehydration in patients with some dehydration as described above.

   Infection Control

   As a routine practice in ICDDR,B hospital the antibiotic treatments for the study children are as follows:

   Children without apparent extraintestinal infection will receive Inj ampicillin @ 100 mg/kg/24 h in 4 divided doses and Inj. gentamicin @ 5mg/kg/24h in 2 divided doses for 5 days. Patients with lower respiratory tract infection will receive Inj: ceftriaxone 75 mg/kg/24 h I/M or I.V one daily doses and Inj. gentamicin 5 mg/kg/24 h in 2 divided doses for 5 days. All patients will receive erythromycin 50 mg/kg/24 h in 4 divided doses for 3 days. Patients with oral thrush will be treated with oral nystacin suspension 100,000 units (1ml) 6 hourly until cured.

   Diet Mother's will be advised to continue breast feeding. Supplementary feeding with F100 diet will be given @ 10 ml/Kg/ Feed two hourly for day 1 and increased slowly up to 150 Kcal/ Kg/Day over 7 days according to the patient's demand. If the child has a poor appetite, or is weak, or has painful stomatitis/glossitis, the food will be introduced through nasogastric tube until the patient will take normal oral feeding. In addition to F100, semisolid food (Rice, lentil, vegetable etc.) will be given to older children during convalescent and rehabilitation phase.

   Vitamin and Mineral Supplements ( As a routine hospital practice in ICDDRB) Children without xeropthalmia and above 1yr of age, will be given vit A 200,000 units and 6-12 months age children will be given 100,000unit on admission. Children with xeropthalmia the same dose will be given on admission, 2nd day and on discharge. Folic acid 1.25 mg and elemental zinc 2 mg/kg will be given for 15 days. In addition children will be given multivitamin supplements (1 ml contains it A palmitate 5000 IU, vitamin D 1000 IU, thiamine hydrochloride 1.6 mg, riboflavin 1 mg, pyridoxine hydrochloride 1 mg, nicotinamide 10 mg, calcium D-pantothenate 5 mg, ascorbic acid 50 mg). 1 ml twice daily for 15 days for 1 yr. and above and half the dose will be given to infants less than <1 yr. of age.

   Hypoglycemia (blood glucose <3 mmol/L) will be managed with 50 ml 10% glucose orally or by nasogastric tube. Hyponatraemia (serum sodium, <115mmol/L with or without symptoms will be managed with Inj. 3% Nacl 12 ml/kg I/V slowly over 4 hrs. Children with serum sodium between 115 - 125 with symptoms will be treated with 3% NaCl in addition to adjunct therapy, if needed.

   Measurements All intakes ( ORS, water, and food) and outputs (stool, urine and vomit) will be measured every 6 hours until diarrhoea stops or upto 7 days . Body weight and vital signs will also be measured 6 hourly.

   Study withdrawal

   Reasons for withdrawal
   1. Any patient developing severe complication such as severe pneumonia, clinical sepsis, meningitis requiring intensive care.
   2. Parents/legal guardian withdraws consent.
   3. Patients who will continue diarrhoea more than 7 days

   Management of withdrawal cases The withdrawal cases will be transferred to general ward or ICU and appropriate management will be provided according to routine hospital practice. Regular follow-up will be done and final outcome of the children will be recorded.

   Data collected up to the time of withdrawal will be included for analysis.

   Management after cessation of diarrhoea ( Convalescent / Rehabilitation Phase) All patients after cessation of diarrhoea and control of other associated infection will be transferred to nutrition rehabilitation unit(NRU) They will be managed with F100 diet according to their requirements. Older children will get semisolid food in addition to F100. During the stay at NRU Vital signs and body weight will be measured once in the morning daily. Food intake will be measured in every feed until the children stay at NRU. After seven days the patients will be discharged from the nutrition rehabilitation unit and will be followed up for next fifteen days at home. They will be supplied with standard diet according to the protocol. The health workers will visit every alternate day and will interview the mother about any illness and approximate amount of diet the child consumed. The health worker will carry a portable electronic balance with a precision of 1 g and record the body weight of the child.

   Definition End of study ( acute phage)- The study end point will be considered when diarrhoea stops or 7 days of initiation of the ORS whichever comes first.

   Cessation of diarrhoea - Diarrhoea will be considered to have stopped when the last watery stool is passed followed by soft or formed stool and/or no stool for 12 hours.

   Hypokalaemia- Hypokalaemia is defined as serum potassium level <3.5 mmol/l. Persistence of hypokalaemia - If the serum potassium level is <3.5 mmol/l on admission and it remains at the level even after 48 hours of therapy with ORS, it will be considered as persistence of hypokalaemia.

   Over hydration - As there are no standard criteria for defining over hydration, we have developed a working definition of over hydration for this protocol based on previous study reports and our clinical experience. Over hydration will be considered in a child who has more than a 5% weight gain than expected after correction of dehydration and / or at least any one of the following signs:

   Development of periorbital oedema; Increased heart rate (>160/min); Increased respiration rate (>60/min); {in the absence of signs suggestive of pneumonia(fever, CXR abnormalities etc.)} Hypoglycaemia - will be defined as blood glucose £ 3 mmol/l

   Hyponatraemia - will be defined as serum sodium < 130 mmol/l

   Severe pneumonia:

   Patient aged 6 m - 12 m

   - respiratory rate > 50/minute with chest in drawing

   Patient aged 13 m - 60 m

   - respiratory rate > 40/minute with chest indrawing (WHO guideline)

   - 'ORS failure' - If after randomization any patient needs I/V rehydration therapy will be labelled as ORS failure.

   Organization of the trial

   Study site - The study will be done in the study ward of the Clinical Service Centre of ICDDR,B.

   Study schedule - The study period will be 2 years from starting.

   Recruiting and training of study personnel - First one month.

   Data collection - 23 months ( Estimated on the basis of bed allotment per protocol and patient availability)

   Data analysis and reporting - 3 months

   OUTCOME VARIABLES

   Primary Duration of diarrhoeal course and stool output.

   Secondary
   1. Calorie intake per day
   2. Daily weight gain
   3. Time to attain 80% weight for height SIGNIFICANCE If the ORS containing amylase resistant starch is found to reduce the severity diarrhoea and increase the recovery in patients with acute diarrhoeal illness in severely malnourished children, it will have a major public health significance as regard to better case management for malnourished children with diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

1. History of acute watery diarrhoea of <72 hrs
2. Either sex
3. Age - 6 months to 60 months
4. Some or severe dehydration
5. Wt for Ht <70% of NCHS median: with or without edema
6. Dark field examination positive for Vibrio cholerae
7. Consent

Exclusion Criteria:

1. Bloody diarrhoea
2. Severe infection (e.g. severe pneumonia, clinical sepsis, meningitis) 3.Those who received antibiotics/antimicrobial for the current illness

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Start 2001-07; Primary Completion 2005-06-30 (Actual); Study Completion 2005-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhoeal course and stool output.

SECONDARY OUTCOMES:
Secondary
Calorie intake per day
Daily weight gain
Time to attain 80% weight for height

CONTACTS AND LOCATIONS:
Overall Officials: Nur H Alam, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh